CLINICAL TRIAL: NCT03989882
Title: Wheat Germ Supplementation Will Improve Markers of Gut Health, Inflammation, and Insulin Resistance in Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS1888
Record Dates: First submitted 2019-05-22; First posted 2019-06-18 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Overweight; Insulin Resistance; Inflammation
Keywords: wheat germ; overweight; gut microbiome; inflammation; insulin resistance
MeSH Terms: conditions — Overweight; Insulin Resistance; Inflammation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know their treatment assignment and energy balls will be in an opaque container.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wheat germ (Experimental): Wheat germ energy balls containing 30 g of wheat germ, peanut butter, and honey to form 2 energy balls that is approximately 200 kcal. Two energy balls will be consumed daily for 30 days.
  Interventions: Other: Wheat germ energy ball
- Control (Placebo Comparator): Control energy ball containing 30 g of cornmeal, peanut butter, and honey to form 2 energy balls that is approximately 200 kcal. Two energy balls will be consumed daily for 30 days.
  Interventions: Other: Control

INTERVENTIONS:
Other: Wheat germ energy ball — wheat germ mixed other ingredients to make an energy ball
  Arms: Wheat germ
Other: Control — corresponding control without wheat germ
  Arms: Control

SUMMARY:
The objective of this pilot study is to determine the effects of wheat germ (WG) supplementation on gut health and subsequent effects on markers of inflammation and insulin resistance in overweight individuals. WG is a by-product of wheat processing and an excellent source of omega-3 fatty acids, vitamin E, and fiber. A few studies have shown the health benefits of WG including gut modulatory potential, but the prebiotic functions of WG in humans remain in question and warrant further investigation.

DETAILED DESCRIPTION:
Healthy overweight (body mass index, BMI, between 25.0 - 30 kg/m2) between 18 to 45 years old regardless of gender will be recruited. They will be randomly assigned to receive two energy balls containing 30 grams of wheat germ or corn meal (control) in a 4-wk randomized controlled pilot trial. The energy balls will contain wheat germ or corn meal, peanut butter, honey and milk. Participants will be asked to consume two energy balls daily for 4 weeks. Anthropometric measures, questionnaires (medical, diet, physical activity and bowel habits), blood and fecal samples will be collected at baseline and at the end of the four week study. The investigator's primary outcome variables will be changes in fecal bacteria, immunoglobulin A, zonulin and short chain fatty acids while secondary outcome variables will be alterations in plasma markers of inflammation and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

Healthy overweight (body mass index, BMI, between 25.0 - 30 kg/m2) 18-45 years old

Exclusion Criteria:

diagnosed diabetes, heart disease, and cancer tobacco use excessive alcohol use taking mega-doses of antioxidant/vitamin supplements or medications that could interfere with study endpoints such as antibiotics, anti-inflammatory, and glucose-lowering medications major surgery occurring within 6 months pregnant or lactating previous high intake of wheat germ or sensitivity to gluten and wheat products.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Fecal bacteria population | Change from baseline fecal bacteria at 30 days
  analyzed by 16sRNA sequencing
Fecal immunoglobulin A | Change from baseline fecal immunoglobulin A at 30 days
  analyzed by enzyme-linked immunoassay
Fecal zonulin | Change from baseline fecal zonulin at 30 days
  analyzed by enzyme-linked immunoassay
Fecal short chain fatty acids | Change from baseline fecal shortchain fatty acids at 30 days
  analyzed by gas chromatography

SECONDARY OUTCOMES:
Blood glucose | Change from baselineblood glucose at 30 days
  analyzed using clinical chemistry analyzer
blood glycated hemoglobin | Change from baseline blood glycated hemoglobin at 30 days
  analyzed using clinical chemistry analyzer
blood high sensitivity C-reactive protein | Change from baseline blood high sensitivity C-reactive protein at 30 days
  analyzed using clinical chemistry analyzer
blood insulin level | Change from baselineblood insulin level at 30 days
  analyzed by enzyme-linked immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Edralin Lucas, PhD, Principal Investigator — Okklahoma State University
Locations (1):
- Nutritional Sciences Department, Oklahoma State University, Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No